CLINICAL TRIAL: NCT07381218
Title: A Prospective, Randomized, and Split-Face Study to Evaluate the Efficacy and Safety of Focused Ultrasound for Facial Skin Laxity
Brief Title: Focused Ultrasound Treatment for Facial Skin Laxity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Huang Lvping, Chief Physician, The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSH-CAMS-HIFU-2025
Record Dates: First submitted 2026-01-13; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Facial Skin Laxity; Skin Aging
Keywords: Focused ultrasound; High-intensity focused ultrasound; Facial skin laxity; Skin aging; Randomized controlled trial; Split-face study

STUDY DESIGN:
Intervention Model Description: This is a randomized split-face study in which each participant serves as their own control. Different focused ultrasound hand-pieces are randomly assigned to opposite sides of the face within the same participant.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Ultrasound with Dot Hand-piece (Experimental)
  Interventions: Device: Focused UltrasoundDot Hand-piece (FUS-D)
- Focused Ultrasound With Micro-focused Hand-piece (Experimental)
  Interventions: Device: Focused Ultrasound Micro-focused Hand-piece (FUS-M)

INTERVENTIONS:
Device: Focused UltrasoundDot Hand-piece (FUS-D) — Focused ultrasound treatment delivered using the dot hand-piece (FUS-D), applied to the contra lateral side of the face during a single treatment session. Treatment parameters follow the predefined study protocol.
  Arms: Focused Ultrasound with Dot Hand-piece
Device: Focused Ultrasound Micro-focused Hand-piece (FUS-M) — Focused ultrasound treatment delivered using the micro-focused hand-piece (FUS-M), applied to one side of the face during a single treatment session. Treatment parameters follow the predefined study protocol.
  Arms: Focused Ultrasound With Micro-focused Hand-piece

SUMMARY:
The goal of this clinical trial is to learn if focused ultrasound can improve facial skin laxity in adults. The main questions this study aims to answer are:

1. Does focused ultrasound treatment lead to clinically meaningful improvement in facial skin laxity compared with baseline assessments?
2. What treatment-related adverse events occur following focused ultrasound treatment, and how frequently and severely do they occur? Researchers will also compare outcomes between the two sides of the face treated with different focused ultrasound hand-pieces within the same participants to explore potential differences in clinical response and safety using a randomized split-face design.

Participants will:

Receive a single session of focused ultrasound treatment applied to both sides of the face.

Undergo standardized clinical assessments, imaging evaluations, and patient-reported outcome measures at baseline and during follow-up visits.

Be monitored for treatment-related adverse events throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Male or female participants
* Presence of mild to moderate facial skin laxity
* Willingness to undergo focused ultrasound treatment of the face
* Ability to understand the study procedures and provide written informed consent
* Willingness to comply with study visits and follow-up assessments

Exclusion Criteria:

* Pregnancy or breastfeeding
* Severe systemic diseases, including but not limited to significant cardiac, hepatic, renal, or neurological disorders
* Active skin infection, inflammation, or open wounds in the treatment area
* History of facial cosmetic procedures (including laser treatment, injectable fillers, or energy-based devices) within the past 6 months
* Presence of implanted electronic devices or metallic implants in the facial area
* Known hypersensitivity or contraindications to focused ultrasound treatment
* Any condition that, in the investigator's judgment, would make the participant unsuitable for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in facial skin laxity from baseline assessed by VISIA skin analysis system | Baseline to 6 months post-treatment
  Facial skin laxity will be quantitatively assessed using the VISIA skin analysis system. Skin laxity-related parameters will be measured at baseline, immediately post-treatment, and at 1, 3, and 6 months post-treatment. Higher values indicate greater skin laxity. The change from baseline at each follow-up time point will be analyzed.
Incidence and severity of treatment-related adverse events | From treatment through 6 months post-treatment
  Treatment-related adverse events will be recorded and evaluated throughout the study, including the type, frequency, and severity of adverse events following focused ultrasound treatment.

SECONDARY OUTCOMES:
Facial skin laxity assessed by VISIA skin analysis system for bilateral facial sides | Baseline to 6 months post-treatment
  Differences in facial skin laxity between the two facial sides treated with different focused ultrasound hand-pieces will be evaluated using the VISIA skin analysis system. Skin laxity-related parameters will be measured at baseline, immediately post-treatment, and at 1, 3, and 6 months post-treatment. Higher values indicate greater skin laxity. A randomized split-face comparison within the same participant will be performed.
Global Aesthetic Improvement Scale (GAIS) score assessed by independent blinded evaluators | From treatment through 6 months post-treatment
  Efficiency of Focused Ultrasound will be assessed using the Global Aesthetic Improvement Scale (GAIS) based on standardized digital facial photographs. GAIS is a 5-point ordinal scale (Grade 1=exceptional improvement; Grade 2=moderate improvement; Grade 3=slight improvement; Grade 4=no change; Grade 5=worsening of the condition). Lower scores indicate better aesthetic improvement. GAIS scores will be measured by both participants and independent blinded evaluators immediately post-treatment, and at 1, 3, and 6 months post-treatment. A randomized split-face comparison within the same participant will be performed.
Wrinkle Severity Rating Scale (WSRS) score assessed by independent blinded evaluators | Baseline to 6 months post-treatment
  Facial wrinkle severity will be assessed using the Wrinkle Severity Rating Scale (WSRS) based on standardized digital facial photographs. WSRS is a validated 5-point ordinal scale (Grade 1=no wrinkles; Grade 2=mild wrinkles; Grade 3=moderate wrinkles; Grade 4=severe wrinkles; Grade 5=very severe wrinkles). Higher scores indicate greater wrinkle severity. WSRS scores will be measured by independent blinded evaluators at baseline, immediately post-treatment, and at 1, 3, and 6 months post-treatment. A randomized split-face comparison within the same participant will be performed.

OTHER OUTCOMES:
Pain intensity score assessed by the Visual Analog Scale (VAS) for bilateral facial sides | Periprocedural
  Pain intensity associated with focused ultrasound treatment will be assessed using the Visual Analog Scale (VAS). VAS is a 10-point scale ranging from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating greater pain intensity. A randomized split-face comparison within the same participant will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Laser Aesthetic Center, Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request, subject to approval by the ethics committee and the study team, and after signing a data use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after study completion and ending 36 months thereafter.
Access Criteria: Data will be shared upon reasonable request, subject to approval by the study team and ethics committee, and after execution of a data use agreement.